CLINICAL TRIAL: NCT04967430
Title: TOGETHER-Toronto: A Phase III Randomized, Double-blind, Placebo-controlled, Multicenter, Trial to Evaluate the Effect of Peginterferon Lambda for the Treatment of COVID-19
Brief Title: TOGETHER - Toronto: Trial to Evaluate the Effect of Peginterferon Lambda for the Treatment of COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JF-12-2020; 21-5018 (Other: University Health Network)
Record Dates: First submitted 2021-07-13; First posted 2021-07-19 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Sars-CoV2; Covid19
Keywords: Peginterferon lambda
MeSH Terms: conditions — COVID-19 | interventions — peginterferon lambda-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): To receive a dose of peginterferon lambda 180mcg SC at baseline (Day 0).
  Interventions: Drug: Peginterferon Lambda-1A
- Placebo (Placebo Comparator): Patients in this arm will receive a single SC dose of 0.9% sodium chloride (normal saline) solution at baseline (Day 0).
  A plastic 1 mL syringe will be prefilled by the study pharmacy. Each syringe will contain 0.5 mL (0.45 mL to match the volume of the Interferon plus 0.05 mL overfill) to allow for needle priming by the unblinded study nurse.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Peginterferon Lambda-1A — Peginterferon lambda is a covalent conjugate of human recombinant non-pegylated IFN lambda (IFN L) and a 20-kDa linear PEG chain.
  Peginterferon lambda Injection is a sterile, nonpyrogenic, ready-to-use solution (0.4 mg/mL) that is clear to opalescent, colorless to pale yellow, and essentially free of particles. Lambda Injection is provided in a 1-mL long Type I glass syringe (0.18 mg/syringe) with a staked 29-gauge, 1/2- inch, thin-walled needle. The syringe has a rigid needle shield and is stoppered with a plunger stopper. Syringes are prefilled with a solution of Peginterferon lambda Injection, mannitol, L-histidine, polysorbate 80, hydrochloric acid, and water for injection; they are intended for a single use at adjustable doses. The syringe is marked with dose indicator lines, which are used as a reference point for administering the correct dose.
  Arms: Treatment
Other: Placebo — The placebo will be 0.9% sodium chloride (normal saline) solution. A plastic 1 mL syringe will be prefilled by the study pharmacy. Each syringe will contain 0.5 mL (0.45 mL to match the volume of the Interferon plus 0.05 mL overfill) to allow for needle priming by the unblinded study nurse.
  Arms: Placebo

SUMMARY:
Interferon (IFN) lambda is one of the fundamental responses of the innate immune system. Peginterferon lambda is a long-acting form that has been studied extensively in human trials in viral hepatitis, confirming it safety and tolerability. It is particularly attractive for consideration in the use of acute respiratory illness due to the high expression of the lambda receptor in lung epithelia. We propose to evaluate peginterferon-lambda in ambulatory patients with mild to moderate COVID-19.

DETAILED DESCRIPTION:
In this study, individuals who attend an Assessment Centre/Emergency Department to be swabbed for COVID-19 and deemed well enough for home isolation will be informed about the study. There will be two major routes of recruitment. Where feasible, a rapid point-of-care (POC) laminar flow based COVID-19 test (the Abbott PanBio) will be performed and those who do not have a POC test at the assessment centre will be tested by PCR.

Interested participants who contact study staff will be confirmed to have a positive COVID-19 test. Once confirmed will be further screened for eligibility criteria by research study staff. After review, a consent form will be emailed to the participant and informed consent will be obtained through witnessed telephone consent from the participant or a substitute decision maker (SDM). Participants who consent will be randomized to receive a single subcutaneous injection of Peginterferon lambda 180µg or saline placebo.

Patients will be followed remotely with visits. In addition, participants will also attend outpatient clinic for swabs and blood work for routine laboratory and inflammatory markers on Days 7 and 14 with the primary endpoint being the time to SARS-CoV-2 RNA negativity and the proportion with COVID-19 related emergency room assessment >6 hours, hospitalization or death by Day 28. Numerous secondary endpoints will be evaluated as well.

Safety data will be reviewed by the Data Safety and Monitoring Committee after the first 50% of randomized participants complete 14 days of follow-up after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18 years of age or older.
2. Symptomatic and within 7 days of symptom onset.
3. High risk for severe disease (as defined by one or more of the following):

   1. Age >50
   2. Diabetes mellitus requiring therapy
   3. Hypertension on medication
   4. BMI >30 kg/m2
   5. Cardiovascular disease
   6. Asthma requiring chronic controller medication
   7. Symptomatic respiratory disease
   8. Immunosuppressed patients (to maximum of 10mg prednisone daily +/- other immunosuppressive agents)
   9. Documented fever (>38C)
   10. One or more of the following symptoms: cough, shortness of breath (SOB), pleuritic chest pain and/or myalgias (to a maximum of 25% of enrollment)
4. Discharged to home isolation.
5. Willing and able to provide informed consent (including by substitute decision maker).
6. Willing and able to follow-up by phone or videoconference.
7. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use adequate methods of contraception during the study and through 90 days after the last dose of study medication. Female patients of childbearing potential are all those except patients who are surgically sterile, who have medically documented ovarian failure, or who are at least 1 year postmenopausal.

Exclusion Criteria:

1. Pregnancy (or positive urine pregnancy test) or lactating.
2. More than 14 days following completion of SARS-CoV-2 vaccition series
3. The following pre-existing medical conditions:

   1. Known cirrhosis with any history of decompensation (ascites, variceal bleeding or hepatic encephalopathy)
   2. Known chronic kidney disease with estimated creatinine clearance < 30 mL/minute or need for dialysis
   3. Uncontrolled severe psychiatric disorder - schizophrenia, bipolar disorder, depression with prior suicidality
   4. Uncontrolled seizures or seizure in the prior 1 month
   5. Any other underlying medical (cardiac, liver, renal, neurological, respiratory) or psychiatric condition that in the view of the investigator would preclude use of peginterferon lambda
4. Known alcohol or drug dependence that in the opinion of the investigator would impair study participation.
5. Known prior intolerance to interferon treatment.
6. Enrolment in another clinical trial testing an antiviral agent or receipt of an antiviral agent for COVID-19 in the past 7 days.
7. Use of investigational, off-label therapy for COVID-19, or unproven therapy for COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 763 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 related urgent care visit, emergency room assessment, hospitalization or death by Day 28 (Primary efficacy endpoint) | At day 28
  Proportion with COVID-19-related emergency room assessment, hospitalization, or death by Day 28
SARS-CoV-2 RNA negativity (Primary virological endpoint) | Day 0 to Day 28
  The time to SARS-CoV-2 RNA negativity.
Treatment-emergent and treatment-related serious adverse events (Primary safety endpoint) | Day 0 to Day 28
  The rate of treatment-emergent and treatment-related serious adverse events (SAEs) by Day 28.

SECONDARY OUTCOMES:
Respiratory symptom resolution (Clinical Outcome #1) | Day 0 to Day 28
  Time to resolution of respiratory symptoms.
Hospitalization (Clinical outcome #2) | Day 0 to Day 28
  Hospitalization for any cause
Death (Clinical outcome #3) | Day 0 to Day 28
  Death due to respiratory or cardiovascular causes
All symptom resolution (Clinical outcome #4) | Day 0 to Day 28
  Time to resolution of all symptoms (return to usual state of heath).
Oxygen saturation on room air (Clinical outcome #5) | Day 0 to Day 14
  Proportion of days with oxygen saturation below 93% on room air by Day 14
Seeking care from healthcare professional for COVID-19 (Clinical outcome #6) | Day 0 - Day 14
  Proportion seeking care from primary care provider/walk-in clinic or study healthcare provider for COVID-19.
Hospital Admission (Clinical outcome #7) | Day 0 to Day 28
  Duration of hospital admission up to Day 28
Time to viral negativity (Virologic/immunological outcome #1) | Day 0 to Day 14
  Time to SARS-CoV-2 RNA negativity.
Mean log of SARS-CoV-2 RNA (Virologic/immunological outcome #2) | Day 3, 5, 7, 10 and 14
  Difference in mean SARS-CoV-2 RNA in log copies/mL
Mean log decline in SARS-CoV-2 RNA (Virologic/immunological outcome #3) | Day 3, 5, 7, 10 and 14
  Difference in mean log decline in SARS-CoV-2 RNA.
Negative for SARS-CoV-2 RNA (Virologic/immunological outcome #4) | Day 3
  Proportion negative for SARS-CoV-2 RNA.
Negative for SARS-CoV-2 RNA (Virologic/immunological outcome #5) | Day 7
  Proportion negative for SARS-CoV-2 RNA.
Negative for SARS-CoV-2 RNA (Virologic/immunological outcome #6) | Day 14
  Proportion negative for SARS-CoV-2 RNA.
Proportion with antibodies (Virologic/immunological outcome #7) | Day 0, 7, 14 and 90
  Proportion with SARS-CoV-2 antibodies in blood.
Correlation with interferon lambda 4 genotype (Virologic/immunological outcome #8) | Day 0 to Day 28
  Correlation of response with interferon lambda 4 (IFNL4) genotype.
Laboratory markers (Virologic/immunological outcome #9) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in hemoglobin over time
Laboratory markers (Virologic/immunological outcome #10) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in white blood cell count over time
Laboratory markers (Virologic/immunological outcome #11) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in lymphocyte count over time.
Laboratory markers (Virologic/immunological outcome #12) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in ALT over time.
Laboratory markers (Virologic/immunological outcome #13) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in AST over time.
Laboratory markers (Virologic/immunological outcome #14) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in ALP over time.
Laboratory markers (Virologic/immunological outcome #15) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in total bilirubin over time.
Inflammatory markers (Virologic/immunological outcome #16) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in lactate dehydrogenase over time.
Inflammatory markers (Virologic/immunological outcome #17) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in c-reactive protein over time.
Inflammatory markers (Virologic/immunological outcome #18) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in D-dimers over time.
Inflammatory markers (Virologic/immunological outcome #19) | Day 0 to Day 7 and Day 7 to Day 14.
  Change in creatine kinase over time.
COVID-19 in household contacts (Transmission outcome #1) | Day 0 to Day 28
  Confirmed diagnosis of COVID-19 in household contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Feld, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No